CLINICAL TRIAL: NCT01740414
Title: Effects of Ibudilast (MN-166, Formerly AV411), a Glial Activation Inhibitor, on Oxycodone Self-administration in Opioid Abusers
Brief Title: Effects of Ibudilast on Oxycodone Self-administration in Opioid Abusers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: #6021; P50DA009236 (NIH)
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Opioid Abuse; Opioid Dependence
Keywords: prescription opioid abuse; pain; opioid withdrawal; oxycodone; ibudilast
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MN-166 (formerly AV411) First (Active Comparator): Participants who began 14-day maintenance on MN-166 (50 mg) first, before switching to Placebo maintenance.
  Interventions: Drug: MN-166 (50 mg) First
- Placebo First (Placebo Comparator): Participants who began 14-day maintenance on Placebo first, before switching to MN-166 (50 mg) maintenance.
  Interventions: Drug: Placebo First

INTERVENTIONS:
Drug: MN-166 (50 mg) First — In this arm of the study participants were first maintained on 50 mg MN-166 BID for approximately 14 days, and were then switched onto placebo maintenance. The subjective and analgesic effects of Oxycodone (0 mg, 15 mg and 30 mg) were tested under each of the two maintenance conditions (Placebo & MN-166).
  Other Names: ibudilast/AV411
  Arms: MN-166 (formerly AV411) First
Drug: Placebo First — This arm of the study participants were first maintained on placebo for approximately 14 days, and were then switched onto 50mg MN-166 BID maintenance. . The subjective and analgesic effects of Oxycodone (0 mg, 15 mg and 30 mg) were tested under each of the two maintenance conditions (Placebo & MN-166).
  Other Names: placebo
  Arms: Placebo First

SUMMARY:
Opioid drugs increase glial cell activation which may be related to the abuse liability of opioid drugs. Data supporting this hypothesis have demonstrated that glial cell attenuators decrease the positive rewarding aspect of opioids in laboratory animals. Ibudilast (MN-166, formerly AV411) is a compound that inhibits the activation of glia. Recent preclinical studies demonstrate that while ibudilast increases the analgesic effects of opioids, it decreases the rewarding effects of such drugs. It has also been shown that ibudilast suppresses morphine-induced release of dopamine, a primary neurotransmitter involved in the rewarding and reinforcing effects of abused drugs. Additionally, we recently found that ibudilast decreases subjective symptoms of opioid withdrawal in opioid dependent humans during detoxification.

Therefore, the primary aim of this 6-7 week inpatient study is to investigate the ability of MN-166 to dose-dependently alter the reinforcing, analgesic, subjective, performance, and physiological effects of oxycodone, a commonly abused prescription opioid.

This study includes a 10-day morphine taper phase, followed by two study phases (approximately 18 days each) with daily active ibudilast and placebo administration, respectively. After the detoxification phase, participants are randomized to receive placebo or MN-166, and then be stabilized on the medication. Thereafter, participants will complete laboratory sessions. Subsequently, during Phase 2, participants will cross over to the other treatment arm, stabilize, and complete laboratory sessions.

DETAILED DESCRIPTION:
Opioid drugs increase glial cell activation and consequent cytokine release. These changes in glial cell activation may be related to the abuse liability of opioid drugs including heroin and prescription opioids. Data supporting this hypothesis have demonstrated that glial cell attenuators decrease the positive rewarding aspect of opioids in laboratory animals. Ibudilast (MN-166, formerly AV411) is a compound that inhibits the activation of glia and thereby inhibits the release of cytokines. Recent preclinical studies demonstrate that while ibudilast increases the analgesic effects of opioids, it decreases the rewarding effects of such drugs. It has also been shown that ibudilast suppresses morphine-induced release of dopamine, a primary neurotransmitter involved in the rewarding and reinforcing effects of abused drugs. Additionally, we recently found that ibudilast decreases subjective symptoms of opioid withdrawal in opioid dependent humans during detoxification.

Therefore, the primary aim of this 6-7 week inpatient study is to investigate the ability of MN-166 to dose-dependently alter the reinforcing, analgesic, subjective, performance, and physiological effects of oxycodone, a commonly abused prescription opioid. A secondary aim is to verify the ability of the drug to decrease opioid withdrawal symptoms during the initial inpatient detoxification.

This inpatient study includes a detoxification and two 18-day study phases. Upon study initiation, participants are tapered with morphine before study phase 1 starts, when they are randomized to receive placebo or 50 mg MN-166 BID (po at 0800 and 2000 hr), and then switched and stabilized on the medication. Thereafter, participants will complete 6 laboratory sessions over 9-10 days.

Subsequently, during Phase 2, participants will cross over to the other study arm (Pbo to MN-166 or MN-166 to Pbo), stabilize, and complete again 6 laboratory sessions. Days 1-10 of the study include a morphine taper, while each of the two subsequent study phases consist of a 7-8-day medication switch and stabilization phase, followed by 6 laboratory sessions over the next 9-10 days (3 sample sessions and 3 choice sessions). During sample sessions, participants will receive one dose of oxycodone (0, 15, or 30 mg/70 kg, PO) that will be available during the choice session the following day. At least 72 hrs after the previous sample session, the second sample session will be completed, followed by a choice session the next day. And then at least 72 hrs after the second sample session, the third and final sample session will be completed, followed by the final choice session the next day. The analgesic, subjective, performance, and physiological effects of oxycodone will be measured. During the choice session, a drug versus money self-administration paradigm will be employed, and the progressive ratio that is completed for drug and/or money will be measured.

We hypothesize that MN-166 will dose-dependently decrease oxycodone self-administration and positive subjective responses while increasing the analgesic effects of the drug.

A secondary additional objective is to collect exploratory information on potential predictors of prescription opioid self-administration including genetic polymorphisms, neurocognitive functioning, and response to stress. Blood samples will be collected to measure various genetic markers hypothesized to contribute to opioid drug effects (e.g., OPRM1, OPRD1, OPRK1, PENK, PDYN, DRD2, CYP3A4, and CYP2D6 genes). Performance on neurocognitive tasks and physiological response to the Trier Social Stress Test will be assessed in all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 21 and 55
* Current opioid dependence according to DSM-IV criteria
* currently not seeking treatment

Exclusion Criteria:

* Female patients that are currently pregnant, or breastfeeding. Lack of effective birth control.
* Participants who have a positive history of neurological illness (including epilepsy) or those who have received anticonvulsant therapy during the past 5 years.
* Liver disease requiring medication or medical treatment, and/or aspartate or alanine aminotransferase levels greater than 3 times the upper limit of normal.
* Gastrointestinal or renal disease that would significantly impair absorption, metabolism or excretion of study drug, or require medication or medical treatment.
* Neurological or psychiatric disorders including psychosis, bipolar disorder, organic brain disease, any seizure history or other disorders that require treatment or that could make study compliance difficult.
* Positive tuberculosis (PPD) TB skin test, clinical history, and chest X-ray indicative of active tuberculosis. (Individuals with a positive PPD test and negative chest X-ray who are not symptomatic for tuberculosis, and do not require antituberculosis therapy will be eligible to participate. Participants will be asked if they ever tested positive for tuberculosis. If so, they will not be given a PPD and chest X-ray and clinical history will be used for evaluation purposes).
* Presence or positive history of severe medical illness or cardiovascular disease or heart abnormality, such as low hemoglobin (Hb < 13 gm/dL in males, Hb < 11 gm/dL in females) with evidence of acute or chronic blood loss, or BP > 140/90.
* Participants on any current psychoactive prescription medications that may interfere with the study measures.
* Current physical dependence on any substance, other than opioids, nicotine or caffeine (ex., methadone, benzodiazepines, LAAM, marijuana, alcohol, etc.).
* Participants for whom detoxification is not "clinically recommended" such as those with a significant history of overdose following detoxification.
* Participation in an investigational drug study within the past 3 months.
* Hypersensitivity to any of the medications used in this study.
* Current (within the last 3 months) chronic pain.
* Platelet and white blood cell count that are not within the normal range (platelet = 120 x103/μl -400 x103/μl; WBC= 3.5 x106/μl -10.8x106/μl).
* Use of Theophylline (PDE-3 inhibitor) or Roflumilast (PDE-4 inhibitor).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — Department of Psychiatry, Columbia University and NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented at conferences and published in peer-reviewed journals.

REFERENCES:
- [Derived] Jacobsen JH, Watkins LR, Hutchinson MR. Discovery of a novel site of opioid action at the innate immune pattern-recognition receptor TLR4 and its role in addiction. Int Rev Neurobiol. 2014;118:129-63. doi: 10.1016/B978-0-12-801284-0.00006-3. PMID 25175864

RESULTS

PARTICIPANT FLOW:
Groups:
- MN-166 First: Patient began maintenance on active medication first (MN-166, formerly AV411) prior to maintenance on placebo.The subjective and analgesic effects of Oxycodone (0 mg, 15 mg and 30 mg) were tested under each of the two maintenance conditions (MN-166, then Placebo).
- Placebo First: Patient began maintenance on placebo medication prior to switching to the active medication condition(MN-166). The subjective and analgesic effects of Oxycodone (0 mg, 15 mg and 30 mg) were tested under each of the two maintenance conditions (Placebo then MN-166).
Period: Overall Study
Arm/Group | MN-166 First | Placebo First
Started | 12 | 16
Completed (This study employed a within-subjects design. Participants completed both MN-166 and Placebo phases.) | 3 | 8
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Population: This was a within-subjects design, however, these numbers denote participant who began with Active (MN-166) maintenance, and those who began under Placebo maintenance.
Groups:
- MN-166 (Formerly AV411): Patient began maintenance on active medication first (MN-166, formerly AV411) prior to maintenance on placebo. The subjective and analgesic effects of Oxycodone (0 mg, 15 mg and 30 mg) were tested under each of the two maintenance conditions (MN-166, then placebo). Data are only from participants who completed both phases of the study.
- Placebo: Patient began maintenance on placebo medication prior to maintenance active medication (MN-166, formerly AV411). The subjective and analgesic effects of Oxycodone (0 mg, 15 mg and 30 mg) were tested under each of the two maintenance conditions (Placebo, then MN-166). Data are only from participants who completed both phases of the study.
- Total: Total of all reporting groups
Arm/Group | MN-166 (Formerly AV411) | Placebo | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (10.8) | 49.5 (1.7) | 42.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Drug Self-administration Breakpoint
Description: Participants are allowed to perform an operant task (click on a mouse) in order to receive a dose drug under investigation (oxycodone dose 0 mg, 15 mg, or 30 mg). The drug breakpoint is the maximum number of responses (mouse clicks) the participant was willing to make to receive the drug. Within the context of abuse liability studies, larger breakpoints represent greater abuse potential of a drug.
Time Frame: 42 days
Measure: Mean (Standard Error); unit: Clicks on a computer mouse
Groups:
- MN-166 + Oxy 0 mg: The Effects of 0 mg of oxycodone while under MN-166 maintenance.
- MN-166 + Oxy 15 mg: The Effects of 15 mg of oxycodone while under MN-166 maintenance.
- MN-166 + Oxy 30 mg: The Effects of 30 mg of oxycodone while under MN-166 maintenance.
- Placebo + Oxy 0 mg: The Effects of 0 mg of oxycodone while under placebo maintenance.
- Placebo + Oxy 15 mg: The Effects of 15 mg of oxycodone while under placebo maintenance.
- Placebo + Oxy 30 mg: The Effects of 30 mg of oxycodone while under placebo maintenance.
Arm/Group | MN-166 + Oxy 0 mg | MN-166 + Oxy 15 mg | MN-166 + Oxy 30 mg | Placebo + Oxy 0 mg | Placebo + Oxy 15 mg | Placebo + Oxy 30 mg
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
Clicks on a computer mouse | 347 (360) | 363 (180) | 1472 (763) | 43 (25) | 1650 (948) | 2459 (1184)

2. Secondary Outcome: Positive Subjective Effects to Oxycodone
Description: Participants are shown a 100-mm line and asked to indicate on that line the extent to which they agree with the descriptor of the drug effect such as "Liking/Liked the Drug." On this visual analog scale participants were instructed that the Left/ 0 mm point on the line represents "not at all," while the right/100 mm point represents "Extremely."
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MN-166 + Oxy 0 mg | MN-166 + Oxy 15 mg | MN-166 + Oxy 30 mg | Placebo + Oxy 0 mg | Placebo + Oxy 15 mg | Placebo + Oxy 30 mg
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
units on a scale | .8 (5.6) | 10.9 (23.9) | 24.2 (35.1) | .9 (3.4) | 15.5 (27.2) | 22.7 (36.9)

3. Other Pre Specified Outcome: Pain Intensity
Description: 15-item shortened form of the McGill Pain Questionnaire (Melzack, 1987) that is used to assess the sensory and affective dimensions of the pain experienced Participants describe their experience of pain by choosing among a series of possible answers (None [score=1], Mild [score=2], Moderate [score=3], or Severe [score=4]). They were asked to describe the pain as "Throbbing," "Shooting," "Stabbing," "Sharp," "Cramping," "Gnawing," "Hot-Burning," "Aching," "Heavy," "Tender," "Splitting," "Tired-Exhausting," "Sickening," "Fearful," and "Punishing-Cruel." Scores were added across all 15 items to generate a sum score, which ranged between 15 and 60.
Time Frame: 42 days
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo Oxy 0 mg: The Effects of 0 mg of oxycodone while under placebo maintenance.
Arm/Group | MN-166 + Oxy 0 mg | MN-166 + Oxy 15 mg | MN-166 + Oxy 30 mg | Placebo Oxy 0 mg | Placebo + Oxy 15 mg | Placebo + Oxy 30 mg
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
units on a scale | 30 (3) | 25 (1) | 26 (2) | 31 (2) | 29 (2) | 27 (2)

ADVERSE EVENTS:
Groups:
- MN-166 (Formerly AV411): Patient is receiving study drug (MN-166) first
  MN-166 (formerly AV411): in one study arm, 50mg MN-166 BID are administered daily for 20 days
- Placebo: Patient is receiving placebo first.
  placebo: In the placebo arm, the patients receive placebo for 20 days
Arm/Group | MN-166 (Formerly AV411) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 3/12 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MN-166 (Formerly AV411) (N=12) | Placebo (N=16)
Insomnia (Nervous system disorders) | 3 (8) | 7 (8)
GI Upset (Gastrointestinal disorders) | 2 (4) | 4 (9)
Headache (Nervous system disorders) | 0 | 2 (3)
Fatigue (Nervous system disorders) | 0 | 2 (5)
Depression (Psychiatric disorders) | 1 (3) | 0
Back Ache (Nervous system disorders) | 0 | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No